CLINICAL TRIAL: NCT00369681
Title: Rituximab and Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Hodgkin's Lymphoma
Brief Title: Phase 2 Study of Rituximab-ABVD in Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0615; P30CA006973 (NIH); NA_00002473 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Rituximab; Dacarbazine; Doxorubicin; Vinblastine

ARMS (1):
- R-ABVD (Experimental): ABVD (doxorubicin; vinblastine; bleomycin; dacarbazine) given as standard for 6-8 cycles. Rituximab given 375 mg/m^2 Cycle 1 Days -6, 1, 8, 15, and 22. Rituximab given 375 mg/m^2 Cycles 2, 4, and 6 Day 1.
  Interventions: Drug: Bleomycin; Biological: Rituximab; Drug: Dacarbazine; Drug: Doxorubicin; Drug: Vinblastine

INTERVENTIONS:
Drug: Bleomycin
  Other Names: Blenoxane
Biological: Rituximab
  Other Names: Rituxan
Drug: Dacarbazine
  Other Names: DTIC; DTIC-Dome
Drug: Doxorubicin
  Other Names: Adriamycin
Drug: Vinblastine
  Other Names: Velban; Alkaban

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating patients with newly diagnosed stage II, stage III, or stage IV Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Investigate plasma DNA biomarkers, including plasma clonal immunoglobulin DNA, tumor suppressor gene methylation, and Epstein-Barr virus DNA, in patients receiving rituximab and doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine (ABVD) for newly diagnosed stage II-IV classical Hodgkin's lymphoma.
* Characterize the impact of rituximab on these markers.
* Characterize the relationship between marker detection and clinical outcome.

Secondary

* Estimate the event-free survival of patients with newly diagnosed Hodgkin's lymphoma treated with rituximab and ABVD.
* Assess the presence of Hodgkin's lymphoma stem cells in peripheral blood mononuclear cells at baseline, after treatment with rituximab, and after treatment with ABVD.
* Assess whether plasma DNA biomarkers add information to fludeoxyglucose F 18 positron emission tomography (FDG-PET) in assessing tumor response.

OUTLINE: Patients receive doxorubicin hydrochloride IV, vinblastine IV, bleomycin IV, and dacarbazine IV (ABVD) on days 1 and 15 of all courses. Patients also receive rituximab IV on days -6, 1, 8, 15, and 22 of ABVD course 1 and on day 1 only of ABVD courses 2, 4, and 6. Treatment repeats every 28 days for 6-8 courses in the absence of disease progression or unacceptable toxicity.

Patients with bulky disease may undergo radiotherapy.

Plasma samples are obtained during treatment for investigation of tumor markers (e.g., immunoglobulin rearrangement, patterns of DNA methylation, and the presence of Epstein-Barr virus DNA). Patients undergo fludeoxyglucose F18 positron emission tomography periodically during the study.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin's lymphoma

  * No lymphocyte-predominant histology
  * Stage II, III, or IV disease
  * Newly diagnosed disease

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Creatinine < 2.0 mg/dL
* Bilirubin < 5 mg/dL
* Not pregnant or nursing
* No HIV positivity
* Hepatitis B surface antigen negative
* No active concurrent malignancy except for superficial nonmelanoma skin cancer or cervical carcinoma in situ

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for Hodgkin's lymphoma
* Steroids allowed if medically required before chemotherapy initiation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L. Kasamon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Background] Kasamon YL, Jacene HA, Gocke CD, Swinnen LJ, Gladstone DE, Perkins B, Link BK, Popplewell LL, Habermann TM, Herman JM, Matsui WH, Jones RJ, Ambinder RF. Phase 2 study of rituximab-ABVD in classical Hodgkin lymphoma. Blood. 2012 May 3;119(18):4129-32. doi: 10.1182/blood-2012-01-402792. Epub 2012 Feb 16. PMID 22343727

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject withdrew consent prior to initiating the study.
Groups:
- R-ABVD: ABVD (Adriamycin/doxorubicin; vinblastine; bleomycin; dacarbazine) given as standard for 6-8 cycles. Rituximab given 375 mg/m^2 Cycle 1 Days -6, 1, 8, 15, and 22. Rituximab given 375 mg/m^2 Cycles 2, 4, and 6 Day 1.
Period: Overall Study
Arm/Group | R-ABVD
Started | 50
Completed | 49
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | R-ABVD
Number analyzed (Participants) | 49
Age, Continuous [Mean (Full Range); unit: years] | 33 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Effect of Rituximab on EBV(+) Tumors
Description: Number of relapses among participants who had tumors positive for Epstein-Barr virus (EBV).
Time Frame: Up to 56 months
Population: Only 4 participants had EBV(+) tumors.
Measure: Number; unit: relapses
Arm/Group | R-ABVD
Number analyzed (Participants) | 4
relapses | 0

2. Primary Outcome: Relationship Between Marker Detection and Clinical Outcome
Description: Number of relapses for participants who did and did not have re-emergence of clonal CD27(+) ALDH(+) B cells after completing study intervention.
Time Frame: 3 years
Population: Only 21 participants had a detectable CD27(+) ALDH(+) clone prior to study intervention. The remaining participants either did not have such a clone or did not have a sample tested to look for a clone.
Measure: Number; unit: relapses
Arm/Group | R-ABVD
Number analyzed (Participants) | 21
relapses
  No re-emergence of clone: number analyzed (Participants) | 16
  No re-emergence of clone | 0
  Re-emergence of clone: number analyzed (Participants) | 5
  Re-emergence of clone | 2

3. Secondary Outcome: Event-free Survival
Description: Percentage of participants who did not experience death, relapse, or progression (worsening) of their lymphoma.
Time Frame: 3 years
Population: All evaluable participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-ABVD
Number analyzed (Participants) | 49
percentage of participants | 83 [68 to 92]

4. Secondary Outcome: Addition of Information to Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) by Plasma DNA Biomarkers
Time Frame: 5 years
Population: Data pertaining to this outcome was not collected.
Arm/Group | R-ABVD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked monthly for up to six months.
Description: Only the following adverse events were collected for this study: all grade 3-5 toxicities; any previously-undescribed toxicity potentially attributable to the addition of the rituximab to the ABVD regimen, regardless of grade; any toxicity associated with infusion of rituximab, regardless of grade.
Arm/Group | R-ABVD
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 16/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-ABVD (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Non-neutropenic infection (Infections and infestations) | 9 (9)
Thrombosis (Vascular disorders) | 4 (4)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Other, not specified (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No